CLINICAL TRIAL: NCT04811066
Title: The Effect of Multi-session Transcranial Direct Current Stimulation Applied Over the Primary Motor Cortex on Motor Sequence Learning in Parkinson's Disease
Brief Title: Motor Learning and Multi-session tDCS in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20200203002
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Transcranial direct current stimulation; Motor sequence learning
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anodal tDCS (Experimental): Anodal electrode (35 cm2 sponge electrode) placed over C3. Cathodal electrode (35 cm2 sponge electrode) placed over the right supraorbital area. 20 minutes of stimulation at 2 mA with a 30-second phase-in and phase-out period.
  Interventions: Device: Transcranial direct current stimulation
- Cathodal tDCS (Experimental): Cathodal electrode (35 cm2 sponge electrode) placed over C3. Anodal electrode (35 cm2 sponge electrode) placed over the right supraorbital area. 20 minutes of stimulation at 2 mA with a 30-second phase-in and phase-out period.
  Interventions: Device: Transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Anodal electrode (35 cm2 sponge electrode) placed over C3. Cathodal electrode (35 cm2 sponge electrode) placed over the right supraorbital area. Stimulation was phased in for 30 seconds up to 2 mA and then switched off. Stimulation was again phased in for 30 seconds following 20 minutes of no stimulation.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial electrical stimulation device. A weak direct electrical current, up to 2 mA, is passed between two electrodes placed on the scalp. Electrodes are housed in 35 cm2 sponges saturated with 4 ml of saline solution (0.9 % NaCl) per side, per pad.
  Stimulation is phased in with a 30-second ramp up of the electrical current to the specified stimulation parameters. Following the specified stimulation period, the current is phased-out with a ramp down of the current. For sham stimulation, the ramp-up and ramp-down periods are retained, but stimulation is switched off during the specified stimulation period.
  Other Names: tDCS

SUMMARY:
The present study seeks to examine the efficacy of multi-session transcranial direct current stimulation applied over the primary motor cortex in people with Parkinson's disease on sequential motor learning performance.

DETAILED DESCRIPTION:
Parkinson's disease is characterised by deficits of motor control triggered by impaired basal ganglia function, such as bradykinesia and tremor. Beyond the visibly recognisable motor symptoms of Parkinson's disease, the ability to learn a sequence of movements is also compromised and poses a significant barrier to effective rehabilitation. In healthy individuals, transcranial direct current stimulation applied over the primary motor cortex during motor task practice has been shown to significantly improve motor learning compared to placebo conditions.

The present study seeks to examine the effect of multi-session transcranial direct current stimulation applied over the primary motor cortex in people with Parkinson's disease on sequential motor learning performance. Participants will be required to attend eight laboratory sessions, comprising five intervention and three assessment sessions and will be tested on their ability to learn a 16-digit finger tapping sequence with their right hand. Sessions one to five will form the intervention and will be performed at the same time on consecutive days (i.e. mon-fri). In addition, session one will double as a baseline assessment and intervention session. Assessments sessions will be performed once before the intervention (session one), and three times following the intervention on day three, one week, and four weeks post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed (Edinburgh Handedness Inventory; ≥50)
* Cognitively capable (Montreal Cognitive Assessment (MoCA); ≥23)
* Mild to moderate Parkinson's disease severity (Hoehn and Yar disease stage 2-3)
* On stable dopaminergic medication

Exclusion Criteria:

* History of stroke
* Comorbidity
* Cephalic implants

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-10-02 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline: sequential finger tapping performance | Four assessments: Baseline (pre-intervention), 3 days, 1 week, and 4 weeks post intervention. Performance is also assessed during the intervention period on each day the intervention is applied. Once immediately before and after intervention is applied.
  A skill index reflecting the accuracy and speed that participants perform a specified finger tapping sequence.
Change from baseline: shape-counting error | Four assessments: Baseline (pre-intervention), 3 days, 1 week, and 4 weeks post intervention. Performance is also assessed during the intervention period on each day the intervention is applied. Once immediately before and after intervention is applied.
  The percentage of shape counting error during dual task assessments. Sequential finger tapping + visual shape counting task.

SECONDARY OUTCOMES:
Change from baseline: oxygenated haemoglobin response | Four assessments: Baseline / pre-intervention, three-days post intervention, 1 week post intervention, and 4 weeks post intervention
  Task related changes of oxygenated haemoglobin as measured using functional near-infrared spectroscopy.
Change from baseline: Movement Disorders Society Unified Parkinson's Disease Rating Scale Motor Section (Part 3) | Four assessments: Baseline / pre-intervention, three-days post intervention, 1 week post intervention, and 4 weeks post intervention
  Participants physical function is assessed according to the criteria of the Movement Disorders Society Unified Parkinson's Disease Rating Scale Motor Section (Part 3). Minimum value = 0, maximum value = 132. Lower scores indicate a better outcome.
Change from baseline: upper limb motor task performance | Four assessments: Baseline / pre-intervention, three-days post intervention, 1 week post intervention, and 4 weeks post intervention
  Timed sequential movement of the arm and hand. The participant sits upright on a chair that has no arm support with their arms relaxed by their side. The time taken to perform the following sequence 10 times is recorded: 1. Close and open hand, 2) flex elbow, 3) close and open hand, 4) extend elbow. Right and left arms are assessed separately.
Change from baseline: Purdue pegboard task performance | Four assessments: Baseline / pre-intervention, three-days post intervention, 1 week post intervention, and 4 weeks post intervention
  Participants are required to pick up a metal peg and place the peg in a specified row of holes. Pegs must be placed one at a time. The maximum number of pegs placed within 30 seconds is recorded. The assessment is repeated three times for each hand. Each hand is assessed separately.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Mak, Dr, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hung Hom, Hong Kong

IPD SHARING:
Plan to Share IPD: No